CLINICAL TRIAL: NCT07317037
Title: ActiTENS Mini (Transcutaneous Electrical Stimulation) in Women With Chronic Pain From Pelvic Endometriosis : a Randomized, Controlled Multicenter Cross-over Study Compared to Weak TENS Treatment, Followed by an Open-label Extension Phase
Brief Title: ActiTENS Mini (Transcutaneous Electrical Stimulation) in Women With Chronic Pain From Pelvic Endometriosis
Acronym: ENDOTENS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: SUBLIMED (Donation of DMs and application development) (Unknown); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: APHP240907; PHRC-23-0046 (Other Grant/Funding Number: Ministry of health, France); 2025-A00238-41 (Other: IDRCB Number)
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Endometriosis
Keywords: pain; endometriosis; trans-cutaneous electrical stimulation; medical device
MeSH Terms: conditions — Endometriosis; Pain

STUDY DESIGN:
Intervention Model Description: A randomized, multicenter, prospective, controlled, cross-over study followed by an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- actiTENS mini - weak stimulation (Other): Adult women suffering from pain related to confirmed pelvic endometriosis, visiting reference and pain centers will be screened for eligibility. If they are eligible and accept to participate (signed informed consent), the DM stimulation mode be assigned by randomization. Patients randomized into this arm will start the study in "actiTENS mini" then "weak stimulation" followed by an open phase where patients can use the DM as they wish.
  Interventions: Device: actiTENS mini - weak stimulation
- weak stimulation - actiTENS mini (Other): Adult women suffering from pain related to confirmed pelvic endometriosis, visiting reference and pain centers will be screened for eligibility. If they are eligible and accept to participate (signed informed consent), the DM stimulation mode be assigned by randomization. Patients randomized into this arm will start the study in "weak stimulation" then "actiTENS mini" followed by an open phase where patients can use the DM as they wish.
  Interventions: Device: weak stimulation - actiTENS mini

INTERVENTIONS:
Device: actiTENS mini - weak stimulation — Patients will wear the DM in "actiTENS mini" mode for 3 months then 1 washout period will be carried out before continuing the study with the DM in mode "weak stimulation" for 3 months. Finally, the last 3-month period will be carried out after 1 month of washout where patients will use the DM as they wish.
  The "weak stimulation" is the control group. The TENS will deliver current for 1 minute every 10 minutes, ramping down to 0 in the last 15 seconds.
  In the experimental group, patients will use the actiTENS mini, which will deliver electrical stimulation: Program P2 (Gate control 80 Hz).
  Arms: actiTENS mini - weak stimulation
Device: weak stimulation - actiTENS mini — Patients will wear the DM in "weak stimulation" mode for 3 months then 1 washout period will be carried out before continuing the study with the DM in mode "actiTENS mini" for 3 months. Finally, the last 3-month period will be carried out after 1 month of washout where patients will use the DM as they wish.
  The "weak stimulation" is the control group. The TENS will deliver current for 1 minute every 10 minutes, ramping down to 0 in the last 15 seconds.
  In the experimental group, patients will use the actiTENS mini, which will deliver electrical stimulation: Program P2 (Gate control 80 Hz).
  Arms: weak stimulation - actiTENS mini

SUMMARY:
Endometriosis is a condition that often causes pelvic pain, particularly during menstruation but also continuously and over long periods. Pharmacological treatments are only moderately effective or are associated with adverse effects. In this context, the search for non-pharmacological approaches to endometriosis pain is essential. Transcutaneous electrical nerve stimulation (TENS) is a portable pain relief technique that is rapidly developing for the treatment of endometriosis pain. The protocol presented aims to confirm the analgesic efficacy of this treatment for endometriosis pain. It will involve 27 gynecology and pain departments in mainland France. It will offer 30-minute sessions of daily stimulation, either suprapubic or lumbar. Several types of stimulation will be compared, with three 3-month phases, two blind phases, and a 3-month phase in which the system used will be fixed. The aim will be to reduce pain intensity as well as other parameters relating to quality of life and the impact of pain. If the effectiveness of this device is confirmed, it could lead to TENS being made available for endometriosis pain and potentially prescribed by gynecologists and midwives.

DETAILED DESCRIPTION:
The study will be proposed to women of adult age during a routine consultation for endometriosis-related pain, in gynecology and pain centers, in France, if they meet the inclusion and exclusion criteria of the study.

Information will be given to them and a necessary period of reflection not exceeding one week will be granted to them.

First phase: a cross-over trial After giving their informed consent, women will be included and randomized either to the actiTENS mini treatment arm or to the low activity treatment arm for 3 months, followed by a wash out period of 28 days. After this first cross-over period, women initially randomized to the actiTENS mini arm will be switched to the low activity arm for 3 months, inversely patients initially in the low activity treatment arm will be switched to the actiTENS mini treatment for the same duration of 3 months.

During the first cross-over study, women will be treated 60 minutes twice daily by a TENS device applied both on the pelvic anterior and sacral posterior region, with the P2 program.

Second phase: an open-label trial After a wash out period of 28 days, all patients will enter the 3-month open phase where only actiTENS mini treatment will be prescribed for 3 months, women choosing freely the region of stimulation (anterior, posterior or both), the program of stimulation and the duration of stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years old
* Followed-up in gynecology consultation for endometriosis confirmed by specific imaging (MRI or ultrasound)
* Referred to a gynecological or a pain center
* With chronic pelvic pain (for at least 3 months) related to endometriosis, pelvic pain being the predominant symptom of endometriosis: pelvic pain present at least 15 days per month in the previous 3 months
* Stable and optimal analgesic and hormonal treatments during the last 3 months: any modification of pharmacological treatment in the last 3 months
* Pelvic pain of moderate to severe intensity or greater than or equal to 4 on an NRS of 0-10 on average during the 8 days preceding the inclusion visit and during the inclusion visit.
* Informed about the concept and accepting the use of TENS as a device, a non-drug analgesic treatment.
* Able to understand the use of TENS
* Having a personal smartphone enabling the EndoTENS application to be downloaded
* All women of childbearing potential (WOCBP) must agree to maintain highly effective contraception by practicing abstinence or by using an effective method of birth control from the date of consent through the end of the study: Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (Oral, Intravaginal, Transdermal); Progestogen-only hormonal contraception associated with inhibition of ovulation (Oral, Injectable, Implantable); Intrauterine device (IUD); Intrauterine hormone-releasing system (IUS); Bilateral tubal occlusion; Vasectomized partner, spermicide-coated condoms
* Willingness and ability to attend the scheduled study visits and comply with study procedures
* Affiliated to Social Security.

Exclusion Criteria:

* Symptoms of endometriosis other than pelvic pain, predominant over pelvic pain (pelvic pain is not the main symptom): digestive disorders, unstable bladder, dyspareunia, infertility, fibromyalgia, sciatica, low back pain…
* Present or past allergy to actiTENS mini pads.
* Pelvic surgery planned within the next 11 months.
* Drug or non-pharmacological treatments not stabilized, which could influence the pathology studied during the last 3 months
* Changed of treatments for endometriosis planned in the next 10 months.
* Patient presenting an absolute contraindication to TENS: patient with epilepsy, patient with a defibrillator, a pacemaker, a cochlear implant or other implanted electronic devices, patient with cardiac disorders, patient with decreased or altered sensation or sensitivity in the area to be treated, for example patients with allodynia (pain triggered by a stimulus that is normally painless) in the area to be treated.
* Patient unable to express his consent or patient in deprivation of liberty.
* Patient that already used or know the functioning principles of a TENS device previously to the clinical study
* Contraindications to actiTENS mini
* Pregnancy and breastfeeding
* Patients under guardianship or curatorship and protected adults
* Patients on AME (Aide Médicale de l'Etat = State Medical Assistance)
* Current participation in another research study involving a therapeutic intervention. Participation to an observational research, or a non-interventional research is allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in the average pain measured with a NRS score of the last 28 days of each 3-month period of treatment, compared to baseline of each period | From the end of the first cross over period (3 months) to the end of the second cross over period (7 months)
  NRS score: 0 is equivalent to no pain and 10 indicates the worst pain.

SECONDARY OUTCOMES:
Efficacy of actiTENS mini on the quality of life | 0 month (baseline for the first crossover period), 1 month, 3 months, 4 months (baseline for the second period), 5 months, 7 months
  Quality of life is measured by EuroQol-5D.
Efficacy of actiTENS mini on the function of patients (EHP-30 and SFSI) | 0 month (baseline for the first cross over period), 1 month, 3 months, 4 months (baseline for the second period), 5 months, 7 months
  Specific functional scores of endometriosis: EHP-30 and SFSI. EHP30 questionnaire is comprised of two parts, the first being the core questionnaire, which consist of five scales (pain, control and powerlessness, emotional wellbeing, social support, and self-image) and contained a total of 30 items. The items within the scales are summed to create a raw score and then each scale was translated into a score ranging from 0 (best health status) to 100 (worst health status)
Efficacy of actiTENS mini on the quality of life and function of patients (PGIC) | 0 month (baseline for the first cross over period), 1 month, 3 months, 4 months (baseline for the second period), 5 months, 7 months
  Global impression of change (PGIC). With this scale, the patient reflects on their perception of the efficacy of the intervention on their limitations regarding activities, symptoms, emotions, and overall quality of life. It consists of a 7-point verbal scale, with the options "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse", and "very much worse"
Number of discharges for ineffectiveness in each group during the 3 months cross-over period | 0 month (baseline for the first cross over period), 1 month, 3 months, 4 months (baseline for the second period), 5 months, 7 months
Better define the analgesic effect of actiTENS mini on endometriosis-related pain by measuring pain using different measures (NRS scale) | 0 month (baseline for the first cross over period), 1 month, 3 months, 4 months (baseline for the second period), 5 months, 7 months
  * Current pain intensity on a NRS from 0 to 10 (0 = no pain and 10 = worst pain imaginable)
  * Background average pain (NRS) over the previous 28 days
  * Pain intensity during flares (NRS)
  * Number of patients with a reduction of 30 and 50% in current pain intensity (NRS)
  * Number of days with pain greater than or equal to 4/10 in the previous 28 days
Better define the analgesic effect of actiTENS mini on endometriosis-related pain by measuring pain (BPI score) | 0 month (baseline for the first cross over period), 1 month, 3 months, 4 months (baseline for the second period), 5 months, 7 months
  Generic functional pain score: BPI score.
Better define the analgesic effect of actiTENS mini on endometriosis-related pain by measuring pain | 0 month (baseline for the first cross over period), 1 month, 3 months, 4 months (baseline for the second period), 5 months, 7 months
  Percentage of Pain Relief since the start of the treatment (% from 0 to 100% of pain relief)
Define the pain profile of responders patients at baseline for actiTENS mini in endometriosis-related pain | 0 month (baseline of the first cross over period), 4 months (baseline of the second period), 8 months (baseline of the third period)
  At the first visit of each phase, a precise evaluation of pelvic pain (location, flares, neuropathic (DN4 questionnaire) and nociplastic component (IASP algorithm for nociplastic pain)), body diagram of pain, and psychological symptoms (HADs questionnaire) of the patients will be carried out, to define the pain phenotypes of patients responding to the treatment (a responder patient is defined as a patient with an average reduction in NRS pain over the last 28 days of 30 to 50% compared to baseline).
Description of the optimal use of actiTENS mini in endometriosis-related pain in routine utilization | 11 months
  During the open-label third phase, at the end (11 months), we will describe the preferred modalities of actiTENS mini use in practice by the patients most of the time (>70%) during this 3-month open label period: TENS programs, TENS electrode location, duration and frequency of stimulation. Quality of life and function questionnaires and measures of pain will also be measured during this third phase.
Comparison of care consumption over the cross-over study periods (Analgesic treatments consumed ) | 0 month (baseline for the first period), 1 month, 3 months, 4 months (baseline for the second period), 5 months, 7 months
  Analgesic treatments consumed since the previous visit at 0, 1, 3, 4, 5, 7 months
Comparison of care consumption over the cross-over study periods (Visits, hospitalizations, emergencies) | 3 months and 7 months
  Visits, hospitalizations, emergencies over the 3 previous months at 3 and 7 months
Device utilization and tolerability of actiTENS mini in the treatment of chronic pain of moderate to severe intensity from endometriosis | 1, 2, 3, 5, 6, 7, 9, 10, 11 months
  Device utilization and tolerability every month through the application by the connected device (type of adverse events and date of occurrence, number of discharges for adverse effects in each group, terms of use of the TENS in case of adverse event).

CONTACTS AND LOCATIONS:
Overall Officials: PERROT Serge, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (27):
- France (27):
  - Chu Amiens Sud, Amiens
  - Clinique Tivoli-Ducos, Bordeaux
  - Chu Cote de Nacre - Caen, Caen
  - Aphp - Antoine Beclere, Clamart
  - Aphp - Louis Mourier, Colombes
  - Chi de Creteil, Créteil
  - Grenoble, Grenoble
  - Aphp - Kremlin Bicetre, Le Kremlin-Bicêtre
  - Hop Jeanne de Flandre Chu Lille, Lille
  - Hopital Croix-Rousse - Hcl, Lyon
  - Hopital Lyon Sud - Hcl, Lyon
  - Aphm - Hopital de La Conception, Marseille
  - Aphm - Hopital Nord, Marseille
  - Chru Nancy - Maternite, Nancy
  - Chu de Nantes Site Hotel Dieu Hme, Nantes
  - Aphp - Pitie Salpetriere, Paris
  - APHP - COCHIN - gynécologie, Paris
  - APHP - COCHIN -centre douleur, Paris
  - GH PARIS SITE SAINT JOSEPH - douleur chronique, Paris
  - Gh Paris Site Saint Joseph, Paris
  - Aphp - Hegp, Paris
  - APHP - Bichat, Paris
  - Chu La Miletrie, Poitiers
  - Ch Rene Dubos - Hopital Novo, Pontoise
  - Hopital Maison Blanche Chu Reims, Reims
  - Chru Rennes Site Hopital Sud, Rennes
  - Chu de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: Yes
The deidentified individual participant data (IPD) that support the results reported in publications may be shared. Additionally, the IPD outlined in the protocol for a planned meta-analysis may also be made available. A data dictionary defining each field will be made available concurrently with the data transmission.
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing requires approval from both the sponsor and the Principal Investigator (PI), contingent upon a scientific project and the PI team's scientific contribution. The founder may also participate in the decision-making process.
  Teams seeking to acquire IPD must engage with the sponsor and the IP team to discuss the scientific (and commercial) objectives, the specific IPD required, the preferred data transmission format, and the proposed timeline. The necessity to inform patients about data sharing or the obligation to undertake procedures with data protection authorities will be evaluated.
  The provision of data through the secure institutional tools of the sponsor AP-HP will be prioritized.
  Technical feasibility and financial support considerations will precede the obligatory formalization of a contract, including detailed description of data processing and general and specific security measures.
  The processing must adhere to the European General Data Protection Regulation.